CLINICAL TRIAL: NCT05315934
Title: A Comparison of the Effects of Upper Versus Lower Body Aerobic Exercise on the Experience of Pain in Individuals With Chronic Knee Pain
Brief Title: Comparing the Effects of Upper and Lower Body Aerobic Exercise on Pain in Individuals With Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Bilzon, Professor James Bilzon, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EP 18/19 088
Record Dates: First submitted 2020-05-17; First posted 2022-04-07 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Chronic Knee Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Body Aerobic Exercise (Experimental): Participants will perform 30 minutes of arm-crank cycling at a moderate exercise intensity based off the participants perceived RPE13
  Interventions: Other: Upper body aerobic exercise
- Lower Body Aerobic Exercise (Experimental): Participants will perform 30 minutes of static cycling at a moderate exercise intensity based off the participants perceived RPE13
  Interventions: Other: Lower body aerobic exercise

INTERVENTIONS:
Other: Upper body aerobic exercise — Participants will perform 30 minutes of continuous exercise on the arm-crank ergometer.
  Arms: Upper Body Aerobic Exercise
Other: Lower body aerobic exercise — Participants will perform 30 minutes of continuous exercise on the cycle ergometer.
  Arms: Lower Body Aerobic Exercise

SUMMARY:
The investigators want to compare the effects of upper versus lower body moderate aerobic exercise on the experience of pain in individuals with chronic knee pain. Participants will attend the laboratory on 4 separate occasions to complete a series of exercise tests and experimental pain tests.

DETAILED DESCRIPTION:
Pain has a multifaceted nature encompassing peripheral drivers (i.e. loading), peripheral and central nervous systems (peripheral and central sensitisation) and cognition (i.e. fear). Most recently, evidence supports that chronic pain in OA may cause alterations to the peripheral and central nervous systems. Despite this, current research has mainly targeted peripheral drivers (usually weight reduction) and cognition (educational programmes) with results highlighting that such methods are not always effective in reducing pain. It would be useful to provide a wider range of choice when prescribing exercise for OA for those which the current prescription is ineffective or un-desirable.

Acutely, both localised and generalised exercise involving the knee joint in individuals with KOA is known to increase symptomatic pain in some. However, research suggests that diverting exercise away from the affected joint may improve pain perception and pain experience in a subset of individuals by targeting cognition (attention away from the joint) and alleviating peripheral drivers of pain (reduced loading) while still presenting systemic physiological benefits that come with acute aerobic exercise which target peripheral and central sensitisation. Currently, there is only one study (Burrows et al, 2014) which has compared the effects of acute upper vs. lower body exercise on pain perception in KOA patients and this was employing resistance exercise. Although this study found positive effects of upper body exercise on pain, this pain was experimentally induced, and symptomatic pain was not measured.

The investigators aim is to determine the effects of a single bout of upper body aerobic exercise on experimentally induced and symptomatic pain in individuals with chronic knee pain in comparison with lower body aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥45 years
* Male or female
* Knee pain for ≥3 months
* Activity related joint pain
* No joint related morning stiffness, or morning stiffness lasting less than 30 minutes.

Exclusion Criteria:

* Specific joint injury within the last 6 months
* Inability to undertake cycling exercise
* Use of anti-inflammatory medication
* Smoker (or having quit <6 months ago)
* Osteoarthritis at any upper body sites that would affect ability to complete arm-cycling exercise.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Acute Symptomatic Pain | Immediately pre and immediately-post exercise
  Change in symptomatic pain measured via Visual Analogue Scale (VAS) from pre- to post-exercise on a 0-10 scale where 0 is no pain at all and 10 is the worst pain imaginable

SECONDARY OUTCOMES:
Acute Experimental Pain | Immediately pre and immediately-post exercise
  Change in experimental pain via Pressure pain threshold and Mechanical detection threshold from pre- to post- exercise
Follow up Symptomatic Pain | 1-7 days post exercise
  Average symptomatic pain in the 7 days following each trial visit measured on a 0-10 Visual Analogue Scale (VAS) where 0 indicates no pain at all and 10 indicates worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymous individual data for all outcomes may be made available.